CLINICAL TRIAL: NCT04984031
Title: Assessment of Apoptosis Markers Caspase-3, Caspase-8, Caspase-9 and Apoptosis Inducing Factor (AIF) Levels in Generalized Versus Molar-incisor Grade C Periodontitis
Brief Title: Apoptosis Markers in Aggressive Periodontitis
Status: Completed | Type: Observational
Sponsor: Asem Mohammed Kamel Ali (Other)
Responsible Party: Sponsor-Investigator, Asem Mohammed Kamel Ali, Principal Investigator, Al-Azhar University
Organization: Al-Azhar University (Other)
Other Study IDs: Apoptosis in periodontitis
Record Dates: First submitted 2021-06-29; First posted 2021-07-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Molar-incisor Pattern Grade C Periodontitis ( Localized Aggressive Periodontitis); Generalized Grade C Periodontitis (Generalized Aggressive Periodontitis)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Generalized grade C periodontitis: generalized aggressive periodontitis ( generalized Grade C ,as in new classification) patients characterized with Bone loss/age index more than 1 and extent more 30 %
  Interventions: Diagnostic Test: ELISA assessment of apoptosis markers in gingival crevicular fluid
- Molar-incisor grade C periodontitis: localized aggressive periodontitis ( Molar-incisor pattern Grade C ,as in new classification) patients characterized with limited affection on molars and incisors and their Bone loss/age index more than 1.
  Interventions: Diagnostic Test: ELISA assessment of apoptosis markers in gingival crevicular fluid

INTERVENTIONS:
Diagnostic Test: ELISA assessment of apoptosis markers in gingival crevicular fluid — Gingival crevicular fluid (GCF) samples will be collected to assess the level of caspase-3,8,9 and apoptosis inducing factor (Aif)

SUMMARY:
The aim of the present trial is to assess the gingival crevicular fluid level of caspase-3 and apoptosis inducing factor (AIF) in Generalized versus Molar-incisor grade C periodontitis.

The present study will be carried out on patients selected from those attending on the outpatient clinics of Department of Oral Medicine, Periodontology, Oral Diagnosis and Dental Radiology, Faculty of Dental Medicine, Al-Azhar University, Assiut.

DETAILED DESCRIPTION:
Periodontal diseases are inflammatory disorders that give rise to tissue damage and loss, as a result of complex interactions between pathogenic bacteria and host immune response. Gingivitis is generally regarded as a site-specific inflammatory condition initiated by dental biofilm accumulation and characterized by gingival redness and edema and the absence of periodontal attachment loss.(1,2) periodontitis, a disease characterized by gingival inflammation combined with connective tissue attachment and bone loss.

Aggressive periodontitis is a form of periodontal disease characterized by rapid attachment loss, bone destruction, non-contributory medical history and family history of the cases Apoptosis is a fundamental and complex biological process that enables an organism to kill and remove unwanted cells during development, normal homeostasis and disease.

Caspases are proteins implicated in the activation and execution of apoptosis was identified in humans as being crucial for this process. Caspases 3 appear to be activated in a protease cascade that leads to inappropriate activation or rapid disablement of key structural proteins and important signaling, homeostatic and repair enzymes and is essential for some of the characteristic changes in cell morphology and certain biochemical events associated with the execution and completion of apoptosis. However, the specific requirements of this caspase in apoptosis were until now largely unknown. Apoptosis-inducing factor (AIF) is a mitochondrion-localized flavoprotein with nicotinamide dinucleotide (NADH) oxidase activity is encoded by a nuclear gene. It has been shown to translocate from mitochondria to the cytosol as well as the nucleus when apoptosis is induced and mediate caspase-independent death because inhibition of caspase activation.

Many authors view apoptosis as a process that is near-to-synonymous to massive caspase activation. The existence of a caspase-independent death effector thus does not fit the dominant scheme. During the last 2 years, several papers advocated the hypothesis that AIF is indeed a caspase-dependent death effector, meaning that the translocation of AIF from the mitochondrion (where it would be inert) to the nucleus (where it would induce apoptosis) would be caspase-dependent.

ELIGIBILITY:
inclusion criteria

1. Patients must be free from any systemic diseases according to criteria of Modified Cornell Medical Index.
2. Males and females aged ≥18 years old.
3. All subjects should be cooperative.

exclusion criteria

1. females, who were lactating or pregnant, will be excluded.
2. smoker's or former smokers also will be excluded .
3. any other periodontal diseases, except generalized grade c periodontitis or molar-incisor grade c periodontitis
4. Patients received antibiotics or non- steroidal anti-inflammatory drugs 3 months or periodontal treatment 6 months' before the beginning of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The present study will carry out on fifty patients ranged in age from (18 - 75) years diagnosed as having aggressive periodontitis. All patients were selected from those attending at outpatient dental clinic of Oral Medicine, Periodontology, Oral Diagnosis and Dental Radiology Department, Faculty of Dental Medicine, Al-Azhar University, Assiut branch. Clinical and radiographic examination will be performed by two calibrated periodontists to confirm accurate diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
caspase 3 , picograms/millimeter (pg/ml) in gingival crevicular fluid | through diagnosis completion, an average of 6 months
  GCF from the mesio-buccal site of each tooth was collected using paper strips held in place for 30 seconds, and then removed. GCF volume (ml) was measured using a calibrated machine. After volume determination, strips were stored in sterile collection tubes that were labeled and then stored at - 80C. Enzyme-linked immunosorbent assays were used to quantify caspase 3 amount in picograms and its concentration (pg/ml) estimated according to the following formula= total caspase 3 amount (pg) / volume GCF (ml).
caspase 8 , picograms/millimeter (pg/ml) in gingival crevicular fluid | through diagnosis completion, an average of 6 months
  GCF from the mesio-buccal site of each tooth was collected using paper strips held in place for 30 seconds, and then removed. GCF volume (ml) was measured using a calibrated machine. After volume determination, strips were stored in sterile collection tubes that were labeled and then stored at - 80C. Enzyme-linked immunosorbent assays were used to quantify caspase 8 amount in picograms and its concentration (pg/ml) estimated according to the following formula= total caspase 8 amount (pg) / volume GCF (ml).
caspase 9 , picograms/millimeter (pg/ml) in gingival crevicular fluid | through diagnosis completion, an average of 6 months
  GCF from the mesio-buccal site of each tooth was collected using paper strips held in place for 30 seconds, and then removed. GCF volume (ml) was measured using a calibrated machine. After volume determination, strips were stored in sterile collection tubes that were labeled and then stored at - 80C. Enzyme-linked immunosorbent assays were used to quantify caspase 9 amount in picograms and its concentration (pg/ml) estimated according to the following formula= total caspase 9 amount (pg) / volume GCF (ml).
Apoptosis Inducing Factor(AIF), picograms/millimeter (pg/ml) in gingival crevicular fluid | through diagnosis completion, an average of 6 months
  GCF from the mesio-buccal site of each tooth was collected using paper strips held in place for 30 seconds, and then removed. GCF volume (ml) was measured using a calibrated machine. After volume determination, strips were stored in sterile collection tubes that were labeled and then stored at - 80C. Enzyme-linked immunosorbent assays were used to quantify AIF amount in picograms and its concentration (pg/ml) estimated according to the following formula= total AIF amount (pg) / volume GCF (ml).

SECONDARY OUTCOMES:
Gingival Index | through diagnosis completion, an average of 6 months
  gingival index used to measure gingival inflammation. The degree of gingival inflammation was assessed as follow: 0 = Normal gingiva.
  1. Mild inflammation, slight change in color, slight edema and no bleeding on probing.
  2. Moderate inflammation, redness, edema and bleeding on probing.
  3. Sever inflammation, marked redness, edema and tendency to spontaneous bleeding.
Plaque Index | through diagnosis completion, an average of 6 months
  Plaque index measured to assess plaque accumulation around gingival margin. The degree of plaque accumulation was assessed as follows:
  0 = no plaque around the gingival margin.
  1. = A thin film of plaque around the gingival margin. The plaque may be recognized only by running a probe across the tooth surface.
  2. = moderate accumulation of soft deposits on the gingival margin and/or adjacent tooth surface, which can be seen by naked eye.
  3. = Abundance plaque accumulation within the gingival pocket and/or on the gingival margin and adjacent tooth surface and hard deposits on the tooth surface are seen.
Attachment level | baseline, immediately after complete diagnosis and before any intervention or therapy
  Attachment level by mm was measured using color -coded probe. The distance from the cemento-enamal junction to the free gingival margin and the distance from the free gingival margin to the base of the pocket where properly measured. The difference between the two measurements yields the attachment level in millimeter (mm).
Bleeding on probing (BOP) | through diagnosis completion, an average of 6 months
  Bleeding on probing (BOP) at a force of 0.3N.with a manual pressure of sensitive probe, recorded on distal, facial, mesial, gingival surfaces.
  Calculation = (Number of bleeding surfaces / total number of tooth surface) *100.Expressed in percentage (%) of gingival units bleeding on probing FMBS.
  In the rating system, 0 indicates absence of bleeding on probing, with 15%, 20% and >20% indicating an increased percentage of inflammation/infection.
radiographic evaluation at molar-incisor area | through diagnosis completion, an average of 6 months
  Marginal bone loss around all central incisors and first molars was evaluated using periapical radiographs. The distance from cemento-enamel junction to the crest of alveolar bone will represent bone lost by mm

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed F Edress, associate professor, Study Director — Faculty of dental medicine Al-Azhar university Assiut Branch; Ahmed M Hussein, phD, Principal Investigator — Oral and Maxillofacial Pathology Department, Faculty of dentistry, Assiut University; Ahmed H Gaber, phD, Principal Investigator — Department of oral pathology Faculty of dental medicine Al-Azhar University (Assiut branch)
Locations (1):
- Faculty of dental medicine Al-Azhar University (Assiut branch), Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gamonal J, Bascones A, Acevedo A, Blanco E, Silva A. Apoptosis in chronic adult periodontitis analyzed by in situ DNA breaks, electron microscopy, and immunohistochemistry. J Periodontol. 2001 Apr;72(4):517-25. doi: 10.1902/jop.2001.72.4.517. PMID 11338305
- [Background] Dabiri D, Halubai S, Layher M, Klausner C, Makhoul H, Lin GH, Eckert G, Abuhussein H, Kamarajan P, Kapila Y. The Role of Apoptotic Factors in Assessing Progression of Periodontal Disease. Int J Dent Oral Sci. 2016 Sep;3(9):318-325. doi: 10.19070/2377-8075-1600064. Epub 2016 Sep 3. PMID 28540365
- [Background] Armitage GC, Cullinan MP. Comparison of the clinical features of chronic and aggressive periodontitis. Periodontol 2000. 2010 Jun;53:12-27. doi: 10.1111/j.1600-0757.2010.00353.x. PMID 20403102
- [Background] Nicholson DW, Thornberry NA. Caspases: killer proteases. Trends Biochem Sci. 1997 Aug;22(8):299-306. doi: 10.1016/s0968-0004(97)01085-2. PMID 9270303